CLINICAL TRIAL: NCT03835923
Title: Lifestyle Intervention in Chronic Ischemic Heart Disease and Diabetes
Acronym: LeIKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Techniker Krankenkasse (Other)
Collaborators: Technical University of Munich (Other); privates Institut für angewandte Versorgungsforschung GmbH (Unknown); IDS Diagnostic Systems AG (Unknown); Federal Joint Committee (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. med. Martin Halle, Univ.-Prof. Dr. med., Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01NVF17015; DRKS00015140 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2019-02-01; First posted 2019-02-11 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Ischemic Heart Disease Chronic; Diabetes Mellitus, Type 2
Keywords: lifestyle intervention; chronic ischemic heart disease; diabetes mellitus type 2; cardiovascular risk factors; health literacy; telemedicine; cross-sectoral care; HbA1c; individual exercise training; dietary change; sustainability; heart disease; nutrition; exercise; physical activity; coronary artery disease; coronary heart disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases; Motor Activity; Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle intervention (Experimental): Telemedicine-supported lifestyle intervention trough individual structured exercise training (endurance and strength training), increase in daily physical activity, and individual nutritional recommendations
  Interventions: Behavioral: lifestyle intervention
- usual care (Active Comparator): general exercise and nutritional recommendations according to current guidelines
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: lifestyle intervention — intervention phase 1 (baseline - month 6): Patients receive an individual exercise plan, nutritional recommendations and advices to increase daily activity. The intervention is accompanied by regular oral and written feedback.
  intervention phase 2 (month 6 - month 12): Patients receive an individual exercise plan, nutritional recommendations and advices to increase daily activity without additional oral or written feedback.
  Arms: lifestyle intervention
Behavioral: usual care — Recommendation for lifestyle intervention at baseline and after 6 months (e.g. salt reduction, restricted alcohol consumption and smoking cessation, 10,000 steps/day, 150 minutes/week moderate intensity exercise)
  Arms: usual care

SUMMARY:
Chronic ischemic heart disease and diabetes mellitus type II have one of the highest morbidity and mortality rates. Especially in the presence of both diseases, these risks increase exponentially. The aim of this program is to reduce cardiovascular risk factors by promoting individual health literacy and a healthy lifestyle, thereby improving metabolism and reducing the progress of the disease as well as mortality.

Patients will receive individual exercise prescriptions and nutritional recommendations. This lifestyle intervention is accompanied by step counters, heart rate sensors, blood glucose meters and smartphones to allow regional implementation in different areas in Germany. In total, 1500 patients with diabetes mellitus type II and chronic ischemic heart disease will participate in the trial.

The project examines whether the intervention positively affects metabolic health and lifestyle behaviors, increases health literacy, and reduces cardiovascular events of these high risk patients. Furthermore, the effectiveness of the intervention will be compared between urban and rural areas.

DETAILED DESCRIPTION:
Chronic ischemic heart disease and diabetes mellitus type II have one of the highest morbidity and mortality rates. Especially in the presence of both diseases, these risks increase exponentially. The combined endpoint of death and myocardial infarction reaches up to 30% within four years. A lifestyle intervention with exercise training and dietary change can reduce the mortality by 20-30% and is a class-I indication in the current guidelines of the European Association of Preventive Cardiology (EAPC). Nevertheless, the implementation of lifestyle interventions in the population is insufficient.

This prospective randomized controlled trial examines whether a structured, individual and telemedicine-supported lifestyle intervention improves health literacy and reduces cardiovascular risk factors compared to a guideline-based recommendation (usual care). Furthermore, the effectiveness of the intervention will be compared between urban and rural areas.

In total, 1500 patients with diabetes mellitus type II and chronic ischemic heart disease will participate in the trial. After randomization (1:1), the 750 patients of the intervention group will receive individual exercise prescriptions and nutritional recommendations based on a maximum exercise stress test and a multi-day nutrition protocol. The intervention is accompanied by pedometers, heart rate sensors, blood glucose meters and smartphones as well as regular oral and written feedback.

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease (ICD-10: I20-I25)
* Diabetes mellitus heart disease (ICD-10: E11)
* insured at participating health insurance
* permission to exercise by the study investigator
* written informed consent

Exclusion Criteria:

* Mental and behavioral disorders (ICD-10: F0-F99)
* Heart failure NYHA IV (ICD-10: I50.14)
* Malignant neoplasm (ICD-10: C25, C34, C56, C72, C73, C78, C79, C97)
* Parkinson's disease (ICD-10: G20)
* Alzheimer's disease (ICD-10: G30)
* infantile cerebral palsy (ICD-10: G80)
* chronic kidney disease (ICD-10: N18.4 & N18.5)
* Trisomy 21 (ICD-10: Q90)
* Blindness / visual impairment (ICD-10: H54.0, H54.2, H54.3)
* Hearing loss (ICD-10: H90.0, H90.3, H90.5, H90.6, H90.8)
* Care level 1-5
* Assured in a foreign country
* Inability to exercise or conditions that may interfere with exercise intervention
* No optimal medical treatment within the last 4 weeks
* Not clinically stable within the last 4 weeks
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  measured in percent (%)

SECONDARY OUTCOMES:
Change in HbA1c | 12 months
  measured in percent (%)
Change in health literacy | 6 and 12 months
  European Health Literacy Survey Questionnaire (HLS-EU-Q16)
Change in daily physical activity | 6 and 12 months
  International Physical Activity Questionnaire (IPAQ)
Change in average steps per day | 6 and 12 months
  7-day average of steps/day measured by pedometers
Change in eating behavior | 6 and 12 months
  Fragebogen zum Essverhalten (FEV; German questionnaire on eating behavior)
Change in quality of life | 6 and 12 months
  Short form health survey (SF-36)
Change of medical care expenses | 6 and 12 months
  routine data of health insurance company
Change in weight | 6 and 12 months
  measured in kilograms (kg)
Change in waist circumference | 6 and 12 months
  measured in centimeters (cm)
Change in LDL-cholesterol concentrations | 6 and 12 months
  measured in milligram/deciliter (mg/dL)
Change in HDL-cholesterol concentrations | 6 and 12 months
  measured in milligram/deciliter (mg/dL)
Change in triglyceride concentrations | 6 and 12 months
  measured in milligram/deciliter (mg/dL)
Change in systolic blood pressure | 6 and 12 months
  measured in millimeters of mercury (mmHG)
Change in diastolic blood pressure | 6 and 12 months
  measured in millimeters of mercury (mmHG)
Number of the combined endpoint "4P-MACE" | 6 and 12 months
  cardiovascular deaths, non-fatal stroke, non-fatal myocardial infarction, hospitalization due to angina pectoris

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, Prof. Dr. med., Principal Investigator — Klinikum rechts der Isar Technische Universität München
Locations (10):
- Germany (10):
  - University Hospital: Rheinisch-Westfälische Technische Hochschule Aachen, Aachen
  - University Hospital: Charité - Universitätsmedizin Berlin, Berlin
  - University Hospital: Herzzentrum Dresden, Dresden
  - University Hospital: Universitäts-Herzzentrum Freiburg - Bad Krozingen, Freiburg im Breisgau
  - University Hospital: Universitätsmedizin Greifswald, Greifswald
  - Doctor's Practice: Dr. Rüdell, Kassel
  - University Hospital: Klinik und Poliklinik für Kardiologie - Universitätsklinikum Leipzig, Leipzig
  - University Hospital: Magdeburg, Magdeburg
  - University Hospital: Klinikum rechts der Isar, Technische Universität München, Munich
  - Doctor's Practice: Prof. Dr. Jacob und Dr. Jacob, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller S, Dinges SMT, Gass F, Fegers-Wustrow I, Treitschke J, von Korn P, Boscheri A, Krotz J, Freigang F, Dubois C, Winzer EB, Linke A, Edelmann F, Feuerstein A, Wolfram O, Schafer K, Verket M, Wolfarth B, Dorr M, Wachter R, Hackenberg B, Rust S, Nebling T, Amelung V, Halle M. Telemedicine-supported lifestyle intervention for glycemic control in patients with CHD and T2DM: multicenter, randomized controlled trial. Nat Med. 2025 Apr;31(4):1203-1213. doi: 10.1038/s41591-025-03498-w. Epub 2025 Feb 7. PMID 39920395
- [Derived] Dinges SM, Krotz J, Gass F, Treitschke J, Fegers-Wustrow I, Geisberger M, Esefeld K, von Korn P, Duvinage A, Edelmann F, Wolfram O, Brandts J, Winzer EB, Wolfarth B, Freigang F, Neubauer S, Nebling T, Hackenberg B, Amelung V, Mueller S, Halle M. Cardiovascular risk factors, exercise capacity and health literacy in patients with chronic ischaemic heart disease and type 2 diabetes mellitus in Germany: Baseline characteristics of the Lifestyle Intervention in Chronic Ischaemic Heart Disease and Type 2 Diabetes study. Diab Vasc Dis Res. 2022 Jul-Aug;19(4):14791641221113781. doi: 10.1177/14791641221113781. PMID 35953083
- [Derived] von Korn P, Sydow H, Neubauer S, Duvinage A, Mocek A, Dinges S, Hackenberg B, Weichenberger M, Schoenfeld J, Amelung V, Mueller S, Halle M. Lifestyle Intervention in Chronic Ischaemic Heart Disease and Type 2 Diabetes (the LeIKD study): study protocol of a prospective, multicentre, randomised, controlled trial. BMJ Open. 2021 Feb 8;11(2):e042818. doi: 10.1136/bmjopen-2020-042818. PMID 33558354